CLINICAL TRIAL: NCT05102357
Title: Retrospective Trial, Scapholunate Ligament Partial Tears in Stable Wrist
Brief Title: Scapholunate Ligament Partial Tears; Tear Localization, Extrinsic Ligament Injury Association and Conservative Treatment Responses Prior to Instability
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Banu Karaalioglu, MD, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: Scapholunate Ligament Tear
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Scapholunate Ligament Partial Tears
Keywords: Scapholunate interosseous ligament, Extrinsic wrist ligaments, Carpal instability, MRI of wrist, Wrist ligamentous injury,
MeSH Terms: interventions — Conservative Treatment; Splints

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Conservative Treatment (splint) — splint 6 weeks

SUMMARY:
The purpose of this study is to investigate scapholunate ligament partial tears regarding tear localization, extrinsic ligament accompaniment in stable wrist and accordingly to scrutinize conservative treatment response.

DETAILED DESCRIPTION:
Patients admitted with radial sided wrist pain without carpal instability were retrospectively evaluated. Scapholunate interosseous ligament (SLIOL) tear localization, grade of injury and associated extrinsic ligament injuries were examined on MRI. Patients treated conservatively and recalled at their first year for re-evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Scapholunate ligament Injury
* Wrist Extrinsic Ligament Injury

Exclusion Criteria:

* Scapholunate Dissociation
* Radiological and clinical instable wrist
* Carpal bone fracture
* MRI imaging artefact

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 109 of 311 patients admitted with radial sided wrist pain had SLL and/or extrinsic ligament injury on MRI, 49,5% (n:55) were female, 50,5% (n:56) male with mean age 34 ± 10 (age range, 12-67 years).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in visual analog scale for pain, disabilities of the arm, shoulder and hand questionnaire and Patient-Rated Wrist Evaluation scores from baseline and at first year | Baseline and 1 year
  Visual analog scale for pain scored from 0 to 10, disabilities of the arm, shoulder and hand questionnaire scored and Patient-Rated Wrist Evaluation scores from from 0 to 100 were scaled at initial admission, before treatment and at their first year recruitment after treatment for assessment conservative treatment success.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kara, Study Director — Medipol University Hospital Department of Orthopedics; Banu Karaalioğlu, Principal Investigator — Medipol University Hospital Department of Radiology
Locations (1):
- Banu Karaalioğlu, Başakşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No